CLINICAL TRIAL: NCT01226576
Title: Focal MR-Guided Focused Ultrasound Treatment of Localized Low-Intermediate Risk Prostate Cancer: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCa004
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Localized Low-Intermediate Risk Prostate Cancer
Keywords: MRgFUS; Prostate Cancer; Low-Intermediate Risk Prostate Cancer; Localized Prostate Cancer; InSightec; ExAblate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): ExAblate Treatment Arm
  Interventions: Device: MRgFUS Treatment

INTERVENTIONS:
Device: MRgFUS Treatment — Local treatment of prostate cancer using Magnetic Resonance Imaging guided endorectally applied focused ultrasound energy
  Other Names: ExAblate 2100 Prostate system

SUMMARY:
The hypothesis of this feasibility study is that focal treatment with ExAblate MRgFUS has the potential to be a safe and effective non-invasive treatment for low to intermediate risk, organ-confined prostate cancer involving low incidence of morbidity. The study hypothesis will be tested by measuring treatment-related safety and initial effectiveness parameters in the ExAblate MRgFUS treated patients, as described above.

Based on the result of this study, InSightec will initiate a larger study in an effort to approve low risk, organ-confined prostate cancer as an indication for its ExAblate MRgFUS device.

DETAILED DESCRIPTION:
Objective of this feasibility trial is to assess safety and initial effectiveness of ExAblate MRgFUS in the treatment of low to intermediate risk, localized (organ confined) prostate cancer tumors.

ExAblate treatment will be implemented as a focal tumor-selective therapy, directed at pre-defined volume(s)/sector(s) in the prostate, (identified as cancerous by mapping biopsy with or without multi-parametric MRI), rather than a whole gland or hemi-ablation treatment.

Safety: evaluate incidence and severity of adverse events associated with ExAblate's MRgFUS focal treatment of low risk organ confined prostate cancer. The risk of ExAblate treatment-related incontinence and impotence will also be assessed in this study.

Effectiveness: determine the tumor control effect of ExAblate's MRgFUS focal treatment of low risk organ-confined prostate cancer (confirmed by TRUS-guided Transperineal Mapping Biopsy results).

ELIGIBILITY:
Inclusion Criteria:

1. Patient of age between 50 to 75 years, inclusive.
2. Biopsy confirmed adenocarcinoma of the prostate, performed up to 6 months prior to scheduled treatment.
3. Patient with low-intermediate risk, early-stage organ-confined prostate cancer (cT1c and cT2a, N0, M0), diagnosed with TRUS guided transperineal biopsy (TPBx) and voluntarily chooses MRgFUS as the non-invasive treatment, who may currently be on watchful waiting or active surveillance and not in need of imminent radical therapy.
4. Patient with PSA less than or equal to 10 ng/mL
5. Gleason score 6 or 7 (no 5 grades), based on TRUS guided Transperineal Mapping Biopsy, as defined in the protocol.
6. Up to two (2) cancerous lesions may be identified in the prostate; each tumor is not more than 10 mm in maximal linear dimension; each tumor should comply with the maximal 7 Gleason score requirement.
7. Positive TRUS-guided transperineal biopsy (TPBx) cores, detected in a maximum of four (4) sectors, (2 for each cancerous focus) out of 16 sectors (or out of 12 sectors in prostates with volume <20 cc)
8. Low grade tumors may or may not be visible by multi-parametric MRI. Thus, in case of MRI-visible tumor, tumor should be in capsular contact of less than 5 mm, on axial images.
9. No definite evidence of extracapsular extension or seminal invasion by MRI
10. Patient eligible for epidural anesthesia, and general anesthesia (in case of complication, requiring intervention).
11. Patient is willing and able to give consent and attend all study visits as defined in the protocol
12. Prostate gland volume should be no greater than 70 cc, volumetrically measured.

Exclusion Criteria:

1. ASA status > 2
2. Contraindications to MRI 2.1. Claustrophobia 2.2. Implanted ferromagnetic materials or foreign objects 2.3. Known intolerance to the MRI contrast agent (e.g. Gadolinium or Magnevist) 2.4. Known contraindication to utilization of MRI contrast agent
3. Severely abnormal coagulation (INR>1.5)
4. Patient with unstable cardiac status including:

   4.1. Unstable angina pectoris on medication 4.2. Documented myocardial infarction within 40 days prior to enrolment 4.3. Congestive heart failure NYHA class IV 4.4. Unstable arrhythmia status, already on anti-arrhythmic drugs
5. Severe hypertension (diastolic BP > 100 on medication)
6. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
7. History of orchiectomy, PCa-specific chemotherapy, cryotherapy, Photodynamic therapy or radical prostatectomy for treatment of prostate cancer; any prior radiation therapy to the pelvis for prostate cancer or any other malignancy.
8. Patient under medications that can affect PSA for the last 3 months prior to MRgFUS treatment (Androgen Deprivation Treatment; alpha reductase inhibitors)
9. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (approximately 3 hrs.)
10. Any rectal pathology, anomaly or previous treatment, which can change acoustic properties of rectal wall or prevent safe probe insertion (e.g., fistula, stenosis, fibrosis).
11. Any spinal pathology which can prevent safe administration of epidural anesthesia
12. Identified calcification of 2 mm or more in largest diameter neighboring the rectal wall (in a distance of less than 5 mm) and interfering with the acoustic beam path.
13. Lower limb musculo-skeletal fixed deformities.
14. Prostate with multiple cystic lesions.
15. Evidence for seminal vesicle/lymph node involvement of cancer.
16. Subjects with distance of the less than 2mm margin between the tumor and the prostate capsule
17. Bladder cancer
18. Patient that had TURP procedure before
19. Urethral stricture/bladder neck contracture
20. Patient with baseline symptoms of incontinence defined as urine leak in any of the following circumstances:

    20.1. Before the patient can get to the toilet 20.2. When coughing or sneezing 20.3. While being asleep 20.4. While being physically active/exercising 20.5. After finishing urinating and being dressed 20.6. Leaking for no obvious reason
21. Patient with baseline impotence scoring 17 or below in the IIEF-5 (SHIM) questionnaire
22. Active UTI
23. Prostatitis NIH categories I, II and III
24. Implant near (<1 cm) the prostate
25. Interest in future fertility
26. Current participation in another clinical investigation of a medical device or a drug or has participated in such a study within 30 days prior to study enrollment

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Safety and initial Effectiveness | 6 months
  1. Safety: incidence and severity of device/treatment related AEs from treatment and up to 6 months follow-up
  2. Evaluating Initial effectiveness of ExAblate MRgFUS to achieve adequate tumor control in low risk organ-confined prostate cancer patients, based on 6-mo Transperineal (TP) mapping biopsy (Bx) findings

SECONDARY OUTCOMES:
Safety | 24 months
  Incidence and severity of device/treatment related AE's from treatment and up to 24 months follow-up
Effectiveness | 24 months
  Evaluating effectiveness of ExAblate MRgFUS to achieve adequate tumor control in low risk organ-confined prostate cancer patients based on periodic PSA follow-up (according to study schedule) and TPBx (Transperineal Biopsy) at two years follow-up. (TPBx will be performed between 6 and 24 months, if clinically indicated)
Effectiveness | 24 months
  Assessing post-ExAblate non-perfused volume (NPV) changes from immediate post- treatment measurement to at 6 and 24 months
QOL | 24 months
  Patients will complete the EPIC-SF12-AUASI questionnaire periodically during study (from baseline up to 24 months post treatment), according to study schedule, to evaluate patient function and satisfaction after prostate cancer treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- University Health Network, Toronto, Ontario, Canada
- Sheba Medical Center, Tel Litwinsky, Israel
- Sapienza University Hospital, Rome, Italy
- National Cancer Center Singapore, Singapore, Singapore
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Lindner U, Ghai S, Spensieri P, Hlasny E, Van Der Kwast TH, McCluskey SA, Haider MA, Kucharczyk W, Trachtenberg J. Focal magnetic resonance guided focused ultrasound for prostate cancer: Initial North American experience. Can Urol Assoc J. 2012 Dec;6(6):E283-6. doi: 10.5489/cuaj.12218. PMID 23283106